CLINICAL TRIAL: NCT06140446
Title: Effect of Two eHealth Applications on Antibiotic Use for Acute, Uncomplicated Upper Respiratory Tract Infections in Children: a Randomized Controlled Trial Among Parents in Dutch General Practice
Brief Title: Effect of eHealth on AB Use of Children With Acute, Uncomplicated URTIs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Max Nieuwdorp (Other)
Responsible Party: Sponsor-Investigator, Max Nieuwdorp, Clinical professor, Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NW2023-49
Record Dates: First submitted 2023-11-14; First posted 2023-11-20 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Upper Respiratory Tract Infection
Keywords: eHealth; Antibiotics; Gut microbiome; General practice
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FeverApp group (Experimental): Use af a self-care FeverApp (containing fever advices and a monitoring function for their child with an uncomplicated URTI), additional to standard advices of the GP.
  Interventions: Device: FeverApp
- DMT group (Experimental): Use of a self-care decision making tool (to choose a herbal medicinal product for their child with an uncomplicated URTI), additional to standard advices from their GP.
  Interventions: Device: DMT App
- Control group (No Intervention): Just standard advices from the GP for their child with an uncomplicated URTI.

INTERVENTIONS:
Device: FeverApp — The (self-management) FeverApp contains evidence-based information about fever and how to deal with it, tailored (phase-oriented) fever advices, and the option to monitor the health status of the child during a fever episode. All information and advices are based on the clinical expertise of paediatricians and the most recent international literature on fever, and complement the Dutch national fever guidelines. It is expected that by letting the body fight the infection on its own in a safe way, less ABs are needed, and the immune system will get stronger leading to less future infections as well.
  Arms: FeverApp group
Device: DMT App — The (self-care) DMT App is a decision making tool (DMT) that can be used by parents to choose a safe and effective herbal medicine (HM) product to reduce symptoms of mild, acute uncomplicated URTIs in their child. The advices that the DMT App provides, are based on a systematic review (SR) of SRs on effectiveness of HM for URTIs, a SR on working mechanisms of the most promising herbs, a prescription rates study of HM for URTIs in 6 European countries, and current EMA status of the included herbs. No prescription from a doctor is needed for these products.
  Arms: DMT group

SUMMARY:
The goal of this clinical trial is to test the effectiveness of two self-care eHealth applications in parents of children with uncomplicated upper respiratory tract infections (URTIs).

The main question it aims to answer is:

• What is the effect of a self-management FeverApp and a self-care herbal medicine decision making tool (DMT) on reducing antibiotic use for acute, uncomplicated URTIs, among children in Dutch general practice?

Participants will:

* Complete an online questionnaire at baseline
* Use a self-care eHealth application for ten days (in the intervention groups)
* Report symptom severity of the URTI of their child online at day 2, 5 an 7
* Complete an online follow-up questionnaire at day 10
* Collect two stool samples of their child at baseline and at day 10

Researchers will compare three groups to see if the Apps have an effect on recovery time and complications from URTIs, AB use, frequency of GP visits, and diversity of the gut microbiome:

* Parents that will use an evidence based fever app additional to standard advices of their GP
* Parents that will use an evidence based herbal medicine DMT additional to standard advices of their GP
* A control group of parents who will receive just standard advices from their GP,

DETAILED DESCRIPTION:
Rationale:

Antimicrobial resistance (AMR) is a complex and growing international public health problem with important consequences as increased mortality and high economic impact. Less inappropriate antibiotic (AB) prescription is one of the global strategies to reduce AMR. In primary care most inappropriate AB prescriptions are for acute, uncomplicated respiratory tract infections (URTIs). URTIs are among the most frequently seen complaints among children in general practice. ABs are only indicated for URTis in case of complications. Nevertheless, they are still often prescribed for uncomplicated cases. A reason for this could be worried parents parents requesting for an AB prescription for their child. In Dutch primary care, ABs can be prescribed by general practitioners (GPs), nurse practitioners (NPs) and physician assistants (PAs). Besides AMR, ABs can cause damage to the gut microbiome. Adequate fever (self) management and safe use of effective (self-care) herbal medicine (HM) are both expected to reduce AB use in mild, acute uncomplicated URTIs. Therefore, a (self-management) FeverApp and a (self-care) herbal medicine decision making tool (DMT App) were developed for parents in general practice.

Objectives:

The primary objective of this study is to investigate the effect of a self-management FeverApp and a self-care DMT App on reducing antibiotic use for acute, uncomplicated URTIs, among children in Dutch general practice. Secondary objectives are to examine (1) amount of apps-related complications and recovery time from acute, uncomplicated URTIs in comparison to standard GP advices, (2) the effect of apps use on reducing the number of GP practice visits and telephone consultations for acute, uncomplicated URTIs, and (3) the effects of apps use (reducing AB use) on diversity of the gut microbiome.

Study design:

The study design is a Randomized Controlled Trial (RCT) in six GP practices. There will be three study groups: (1) a group of parents who will be advised to use the FeverApp additional to advices from their GP practice, (2) a group of parents who will be advised to use the self-care DMT App additional to advices from their GP practice, and (3) a control group of parents who will only receive advices from their GP practice. Recruitment of parents will be done by the GP practice assistants of the participating practices, and selection and inclusion will be carried out by a research assistant from University of Applied Sciences Leiden (UAS Leiden). Randomization over the conditions will be done at random by the research assistant. This will result in parents assigned to either the Fever App group, the DMT App group or the control group. All included parents will, after receiving the participant information, fill out a baseline online questionnaire (including digital informed consent), and will collect a baseline stool sample of their child and save it in the freezer (T0). After that, parents in the intervention groups download and use the app they were assigned to, and all parents report (severity of) URTI symptoms of their child online at 2, 5 and 7 days (T1, T2 and T3) in an online form. Ten days after T0, all parents fill out a follow-up questionnaire, collect a second stool sample from their child, and save it in their own -20 degrees Celsius freezer (T4). At the end of the study, all of the stool samples will be picked up at home by research assistants from UAS Leiden, and will be transferred to Amsterdam University Medical Centre for the laboratory gut microbiome analysis.

Benefits, burden and risks:

The benefit of participating in the study, is that parents in the intervention groups will get extra support by means of the apps, on top of the advices that will be provided by the GP practice. For the control group there is no real benefit, besides contributing to less AB use among children in the future. The burden of this study lies in the fact that parents who participate, will have to fill out two online questionnaires within two weeks, report symptom severity online at two more timepoints, and will have to collect a stool sample of their child twice and save it in the freezer. Parents in the intervention groups will get the advice to download and use one of the two investigated apps. It will be their own decision to actually do this or not.

Participating in the study is safe, because only parents of children with mild, acute, uncomplicated URTIs will be involved. Furthermore, advices/care by the GP practice will be continued for all patients in the study, and the advices in the (self-management) fever app are in line with national fever guidelines. The only difference is that, based on the most recent insights on fever, the app encourages to keep the child warm in the first phase of fever. With regards to safety of the (self-care) DMT App, adverse events due to HM are rare. Moreover, the herbs that are advised on in the app are freely available (without prescription) in drugstores and pharmacies in the Netherlands. Therefore, using the (self-care) DMT App will make things safer rather than less safe, because parents in the HM group will get a trustworthy advice based on scientific evidence and safety regulations, instead of buying herbal medicine without an evidence-based decision-making tool (DMT) like they would normally do.

All participating parents will be advised to always go to the national website with GP advices in case of doubts about the health status of their child, and to call their GP practice, the ED (emergency department) or 112 in case of alarm symptoms. Furthermore, all parents are told to report complications from the URTI and/or adverse events (such as hospitalization) to the researchers. In case of complications or adverse events, they will be will go back to just receiving advices/care from their GP/NP/PA. Participating parents will use the apps in a test account, so no data will be collected by the apps. Also, the online questionnaires they fill out are anonymous, so the privacy of parents who participate is secured. Finally, parents can leave the study at any moment and go back to just receiving advices from their GP practice. There is no relation between (parents in) the different study groups.

ELIGIBILITY:
Inclusion Criteria:

* Having a child aged 0-12 years old
* Master the Dutch language
* Having called the GP for their child aged 0-12 years having:

  * Fever (≥38 °C) AND
  * At least one of the following symptoms:

    * Acute cough
    * Sore throat
    * Earache/runny ear
    * Nasal congestion/runny nose
    * Headache
* Being screened by a triage specialist (GP practice assistant) and not being indicated for a GP/NP/PA visit
* Not being included in the trial before

Exclusion Criteria:

* The current URTI complaints of the child already exist longer than 2 weeks
* The child who has a URTI

  * is younger than 3 months old
  * has asthma or another chronic or severe illness
  * has a history of pneumonia
  * has a history of complications or hospitalization from a previous URTI
  * has Down Syndrome
  * has a less functioning immune system
* The parent being very worried

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 411 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Antibiotic use (yes/no) | Self-reported10 days after inclusion in the study
  Antibiotic use of the child in the current URTI episode

SECONDARY OUTCOMES:
Normal recovery time from URTI | Self-reported 10 days after inclusion in the study
  Recovery of the URTI within 7 days (based on the clinical expertise of GPs)
Adverse events/complications | Self-reported 10 days after inclusion in the study
  Adverse events/complications from current URTI
GP visits | Self-reported 10 days after inclusion in the study
  Number of follow-up GP/NP/PA visits for the current URTI episode
Telephone consultations | Self-reported 10 days after inclusion in the study
  Number of follow-up telephone consultations for the current URTI episode of the child
Gut microbiome diversity | At baseline (inclusion) AND 10 days after inclusion in the study
  Change in diversity of the gut microbiome (by means of stool samples)
AB type | Self-reported at 10 days after inclusion in the study
  Type of AB used in current URTI episode
AB dosage | Self-reported at 10 days after inclusion in the study
  AB dosage used in current URTI episode

CONTACTS AND LOCATIONS:
Overall Officials: Max Nieuwdorp, PhD, Study Director — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam UMC location AMC, Amsterdam, Netherlands

REFERENCES:
- [Derived] Belt-van Zoen E, van Steenbergen N, Veldman L, Nieuwdorp M, Baars EW. Evaluating the effects of two parental self-management eHealth applications on antibiotic use, number of primary care visits and gut microbiota of febrile Dutch children with acute, uncomplicated upper respiratory tract infections: a study protocol for a randomised controlled trial. BMJ Open. 2025 Dec 19;15(12):e101463. doi: 10.1136/bmjopen-2025-101463. PMID 41419287